CLINICAL TRIAL: NCT03285035
Title: Quality of Life Assessment in Patients Receiving Cryotherapy in Addition to Chemotherapy for Palliation of Unresectable Esophageal or Gastroesophageal Cancer
Brief Title: Quality of Life Assessment of Cryotherapy in Esophageal or Gastroesophageal Cancer
Acronym: Cryotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: WG2015029
Record Dates: First submitted 2017-08-28; First posted 2017-09-15 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Esophageal Cancer
Keywords: Cryotherapy; Palliation; Dysphagia
MeSH Terms: conditions — Esophageal Neoplasms; Deglutition Disorders | interventions — Cryotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archival tissue or fresh tissue from gastrointestinal biopsies used for diagnostic purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Non-operable esophageal cancer: Cryotherapy treatment
  Interventions: Device: Administration of questionaires to patients receiving an upper endoscopy with cryotherapy in addition to chemotherapy for esophageal cancer palliation.

INTERVENTIONS:
Device: Administration of questionaires to patients receiving an upper endoscopy with cryotherapy in addition to chemotherapy for esophageal cancer palliation. — Upper endoscopy with cryotherapy using liquid nitrogen.

SUMMARY:
Cryoablation combined with chemotherapy on the quality of life of patients with non resectable esophageal or gastroesophageal cancer.

DETAILED DESCRIPTION:
This is a single arm prospective study to determine the effect of cryoablation combined with chemotherapy on the quality of life of patients with non resectable esophageal or gastroesophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has esophageal or gastroesophageal cancer and will be receiving chemotherapy
* Dysphagia score of 1, 2, 3 or 4.
* Age ≥18 years old
* American Society of Anesthesiologists (ASA) Physical Status Classification ≤ 4
* Deemed not a candidate for esophageal cancer surgical resection
* Female subjects must be either post-menopausal, surgically sterilized, or willing to use an acceptable method of birth control (i.e., total abstinence, birth control pills, an intrauterine device (IUD), diaphragm, progesterone injections or implants, or condoms plus a spermicide) for the duration of the study

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status greater than 2
* Patient who received radiation treatment in the prior 8 weeks
* Known brain metastases causing cranial nerve deficits which can cause dysphagia
* Inability to undergo an esophagogastroduodenoscopy (EGD)
* Pregnant or nursing
* Surgery or anatomy where capacity of stomach is reduced making cryotherapy contraindicated
* Patients with tracheoesophageal fistula

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with non resectable esophageal cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-07-13 (Actual); Primary Completion 2020-07-13 (Estimated); Study Completion 2021-01-13 (Estimated)

PRIMARY OUTCOMES:
Change in baseline quality of life (QOL) assessment using a modified EORTC QLQ-OES18 at 6 months compared to baseline | 6 months

SECONDARY OUTCOMES:
Change in dysphagia score using the 5 point Likert scale at 1 to 2 weeks post-procedure compared to baseline | 1 to 2 weeks
Number of participants with adverse events as assessed by CTCAE 4.03. | 30 days
Number of participants requiring alternative treatments for dysphagia palliation such as stenting, photodynamic therapy or brachytherapy and stenting | 1 year
Subjective Global Assessment scale of nutritonal status will be determined at baseline and approximately 3 month intervals. | 1 year
Tumor length in centimeters, endoscopist estimated luminal diameter and endoscopist subjective assessment of size as compared to the prior endoscopy will be determined | 1 to 12 weeks
Immunoassays will be obtained before and after treatment | 1 year
local tumor control will be compared to systemic tumor control | 1 year
Survival while on cryotherapy and systemic chemotherapy will be measured. | 1 year
Change in baseline quality of life (QOL) assessment using a modified EORTC QLQ-OES18 at 1 to 2 weeks compared to baseline | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Toufic Kachaamy, MD, Principal Investigator — Western Regional Medical Center
Locations (1):
- Western Regional Medical Center, Inc., Goodyear, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kachaamy T, Sharma N, Shah T, Mohapatra S, Pollard K, Zelt C, Jewett E, Garcia R, Munsey R, Gupta S, Rojas-DeLeon M, Gupta D, Kaul V, Pannala R, Vashi P. A prospective multicenter study to evaluate the impact of cryotherapy on dysphagia and quality of life in patients with inoperable esophageal cancer. Endoscopy. 2023 Oct;55(10):889-897. doi: 10.1055/a-2105-2177. Epub 2023 Jun 2. PMID 37268010